CLINICAL TRIAL: NCT03227003
Title: Dietary Intake of One-carbon Metabolism Nutrients and DNA Methylation in Peripheral Blood
Brief Title: DNA Methylation and 1-C Metabolism Nutrient Intake
Status: Completed | Type: Observational
Sponsor: Cancer Council Victoria (Other)
Responsible Party: Principal Investigator, Roger Milne, Head, Cancer Epidemiology & Intelligence Division, Cancer Council Victoria
Other Study IDs: CEID_methylation_1
Record Dates: First submitted 2017-07-21; First posted 2017-07-24 (Actual); Last update posted 2017-07-24 (Actual); Status verified 2017-07

CONDITIONS: DNA Methylation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The present study used a sub-sample of the Melbourne Collaborative Cohort Study (MCCS) (Milne RL et al, Int J Epidemiol, 2017), who had valid data on dietary intakes (121-item food frequency questionnaire) and valid measures of DNA methylation using the HumanMethylation Infinium 450K Beadchip assay, or using LINE-1, Alu and Sat2 assays.

The investigators studied the association between nutrients involved in one-carbon metabolism and DNA methylation in peripheral blood.

ELIGIBILITY:
Inclusion Criteria:

* Selected into one of six case-control studies nested in the Melbourne Collaborative Cohort Study
* Completed a 121-item Food Frequency Questionnaire
* Had a blood DNA sample with a measure of methylation

Exclusion Criteria:

* Missing data in any of the outcome, exposure, or confounders (N=797 excluded)

Ages: 27 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population is a sub-sample of the Melbourne Collaborative Cohort Study (MCCS), with non-random sampling based on selection into of six case-control studies nested within the MCCS. The MCCS is a prospective cohort study of 41,513 people (17,044 men and 24,469 women) recruited between 1990 and 1994. The age range at recruitment was 27-80 (99.3% being aged 40-69). Southern European migrants to Australia were over-sampled to extend the range of exposures, including dietary patterns.
  Participants in this sub-study had valid dietary intake data and valid measures of DNA methylation.
Sampling Method: Non-Probability Sample
Enrollment: 5983 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Blood DNA methylation | 2014-2015
  Methylation of DNA from peripheral blood, HumanMethylation 450 Beadchip assay

SECONDARY OUTCOMES:
Blood DNA methylation | 2014-2015
  Methylation of DNA from peripheral blood, LINE-1, Alu, Sat2

CONTACTS AND LOCATIONS:
Overall Officials: Graham G Giles, PhD, Principal Investigator — Cancer Council Victoria

REFERENCES:
- [Derived] Chamberlain JA, Dugue PA, Bassett JK, Hodge AM, Brinkman MT, Joo JE, Jung CH, Makalic E, Schmidt DF, Hopper JL, Buchanan DD, English DR, Southey MC, Giles GG, Milne RL. Dietary intake of one-carbon metabolism nutrients and DNA methylation in peripheral blood. Am J Clin Nutr. 2018 Sep 1;108(3):611-621. doi: 10.1093/ajcn/nqy119. PMID 30101351